CLINICAL TRIAL: NCT04187638
Title: Effect of Olive Oil Consumption on Cardiovascular Biomarkers in Asians and Caucasians: A Randomized, Crossover, Controlled Interventional Trial
Brief Title: Effect of Olive Oil Consumption on Cardiovascular Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Jose Lara Gallegos, Senior Lecturer, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HLS-JLG-OOstudy
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Olive Oil; Butter

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled crossover trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil (Experimental): Participants will receive 30ml/day of olive oil for two weeks
  Interventions: Dietary Supplement: Olive oil; Dietary Supplement: Butter
- Butter (Placebo Comparator): Participants will receive 30g/day of butter also for two weeks.
  Interventions: Dietary Supplement: Olive oil; Dietary Supplement: Butter

INTERVENTIONS:
Dietary Supplement: Olive oil — Participants will be randomly allocated to receive daily dose of 30ml of olive oil (OO) as intervention group or a matching control (butter 30g) for 2 weeks each (i.e. two weeks olive oil and two weeks butter), separated by a washout period of 2 weeks between treatments.
Dietary Supplement: Butter — Participants will be randomly allocated to receive daily dose of 30ml of olive oil (OO) as intervention group or a matching control (butter 30g) for 2 weeks each (i.e. two weeks olive oil and two weeks butter), separated by a washout period of 2 weeks between treatments.

SUMMARY:
The main aim of this study is to examine the effect of olive oil consumption on several cardiovascular risk markers between Caucasians and Asian ethnicity. The primary assessments: endothelial function's biomarkers: cell and vascular adhesion molecules (ICAMs and VCAMs) and nitric oxide (NO). The secondary assessments: Lipid profile.

ELIGIBILITY:
Inclusion Criteria:

Male

Orient Asians (including Chinese, Japanese, Korean, and Malaysia Chinese) and Caucasians

Age 18-70 years

Self-reported in good general health

Exclusion Criteria:

Female

Age older than 70 years or younger than 18 years

Diagnosed and/or are taking medications for hypertension (>140/90mmHg)

Diabetes

High blood cholesterol

Heart problems (e.g. arrhythmia, high-grade stenosis of the carotid artery or carotid sinus syndrome)

Allergy to olive oil or olive oil products

Lactose intolerance

Taking omega-3 supplements in fish oil and vitamins supplements in the last six months.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
changes in ambulatory blood pressure | Baseline and 2 weeks

SECONDARY OUTCOMES:
Changes in plasma total cholesterol | Baseline and 2 weeks
  Plasma total cholesterol vascular cell adhesion molecule 1
Changes in Intercellular Adhesion Molecule 1 | Baseline and 2 weeks
  Plasma levels of Intercellular Adhesion Molecule 1 measured
Changes in vascular cell adhesion molecule 1 | Baseline and 2 weeks
  Plasma levels of vascular cell adhesion molecule 1 measured
Changes in C-reactive protein | Baseline and 2 weeks
  Plasma levels of CRP measured

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Applied Sciences, Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No